CLINICAL TRIAL: NCT02751580
Title: TELEPORT STUDY: A Pilot Feasibility Trial Examining The Use of Telehealth in Post Radiation Therapy Visits
Brief Title: Telehealth in Improving Quality of Life in Patients During Post Radiation Therapy Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15D.580; JT 8256 (Other: JeffTrial Number)
Record Dates: First submitted 2016-04-11; First posted 2016-04-26 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Health services research (telehealth) (Experimental): Patients undergo their first post-treatment visit as a virtual telehealth visit using the JeffConnect application downloaded onto their electronic device.
  Interventions: Other: Telemedicine; Other: Questionnaire Administration

INTERVENTIONS:
Other: Telemedicine — Attend a virtual visit via the JeffConnect telehealth app
  Other Names: Telehealth
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well telehealth works in patients during post radiation therapy visits. A telehealth virtual office visit can be performed from the patient's home or workplace, decreasing time spent traveling to visit site, time spent in waiting room, and cost to patient. Studying telehealth may improve quality of life in patients during post radiation therapy visit.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine feasibility of conducting a trial comparing a telehealth visit and an in person office visit.

SECONDARY OBJECTIVES:

I. To examine patient satisfaction, patient assessment of physician communication during a telehealth visit.

II. To examine patient distrust in the healthcare system following a telehealth visit.

III. To examine physician ability to perform a patient assessment during a telehealth visit.

IV. To examine physician perceptions of telehealth visits. V. To examine monetary and time cost to patients for telehealth visit. VI. To calculate clinic savings derived from telehealth visits.

OUTLINE:

Patients undergo their first post-treatment visit as a virtual telehealth visit using the JeffConnect application.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently undergoing or planned to start radiation treatment with curative, adjuvant or palliative intent
* Karnofsky performance status (KPS) score >= 60
* Patients must be capable to read and speak English and provide study specific informed consent prior to study entry
* Patients must have access to a computer or smartphone and internet connection at home on which they would be willing to do a telehealth study
* Pennsylvania or New Jersey residents *Telehealth visits for New Jersey residents will only be performed by physicians with a current medical license issued by the state of New Jersey.

Exclusion Criteria:

* KPS < 60%
* No access to a computer, smartphone or internet
* Unable to read and/or speak English
* Decisionally impaired patients
* Patients not residing in Pennsylvania or New Jersey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Simone, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Services Research (Telehealth)
Started | 37
Completed | 31
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Conducting a Future Randomized Clinical Trial Comparing Telehealth and in Person Visits (i.e., Rate of Accrual)
Description: The number of patients accrued each month will be analyzed via Poisson regression. The mean (monthly rate) will be estimated and tested against the null value of 4 patients per month using a 1-sided test with alpha 0.05. The proportion of enrolled subjects who are lost to follow-up will also be summarized.
Time Frame: 24 months from first patient enrolled
Population: 13 participants did not complete the Telehealth visit: 7 did not show for their appointment, 4 were never scheduled, 1 patient passed away prior to completion of visit and 1 patient canceled the appointment in favor of hospice care
Measure: Mean (Standard Deviation); unit: participants accrued per month
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 37
participants accrued per month | 2.4 (1.67)

2. Secondary Outcome: Patient Satisfaction With Telehealth Visits as Measured by the Patients Satisfaction With Cancer Care Score
Description: Patients Satisfaction with Cancer Care score is an 18-item questionnaire with answers on a 5-point Likert scale. Lower scores are associated with higher satisfaction with caner care. The average will be computed and tested against the null value of 75 using a one-sample t-test with alpha 0.05.
Time Frame: 4 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 37
Participants
  Strongly agreed | 32
  Agreed | 5

3. Secondary Outcome: Number of Patients Satisfied With Physician Communication During Telehealth Visit
Description: 14 item communication assessment tool (CAT). The CAT addresses specifically patient satisfaction with key aspects of communication and interpersonal skills and items are scored on a 1-5 scale where 1 = poor and 5 = excellent and a higher score would indicate better communication skills
Time Frame: 4 months from enrollment
Population: All 37 patients analyzed report satisfaction
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 37
Participants | 37

4. Secondary Outcome: Patient Distrust in the Healthcare System as Measured by the Health Care System Distrust Scale in Relation to Privacy of Medical Record (MR)
Description: healthcare system distrust scale, designed to assess the belief that physicians would act in a patient's best interest to prevent a potentially negative important outcome (ref). This is a 10 item survey scored 1-5 where 1 = "strongly disagree" and 5 = "strongly agree" and higher scores generally indicate more distrust. Patient distrust was measured by asking if patients felt their Medical Record (MR) would be kept private or would be accessed without their permission.
Time Frame: 4 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 37
Participants
  Agree MR could be access without permission | 5
  Unsure MR are kept private | 5

5. Secondary Outcome: Physicians Ability to Evaluate a Patient During a Telehealth Visit as Measured by the Physician Questionnaire
Description: 9 question survey regarding the ease of use and efficacy of the telehealth platform. The items were yes or no questions (scored on 1 = yes and 0 = no) scale. Higher scores represent greater satisfaction with the platform.
Time Frame: 4 months from enrollment
Population: 9 physicians and 2 nurses evaluated the use of telehealth platform
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 11
Participants
  Assess Symptoms | 11
  Assess Treatment-Related Toxicity | 9

6. Secondary Outcome: Physician Satisfaction With Post-treatment Telehealth Visit as Measured by the Modified Physician Satisfaction Scale
Description: 9-question survey regarding the ease of use and efficacy of the telehealth platform. The items were yes or no questions (scored on 1=yes and 0=no) scale. Higher scores represented greater satisfaction with the platform. Specifically looked at responses to the items regarding: accurate assessment of symptoms via telehealth, accurately assess treatment-related toxicity via telehealth, feeling sure they obtained all information needed to care for the patient, and if providers would use the telehealth system in the future.
Time Frame: 4 months from enrollment
Population: 9 physicians and 2 nurse practitioners
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 11
Participants
  Accurately Assess Symptoms | 11
  Accurately Assess Treatment-related toxicity | 9
  Obtained All Information Needed for Patient Care | 8
  Agreed Would Use Telehealth in future | 10

7. Secondary Outcome: Patient Costs for Telehealth Visit
Description: Patient costs for telehealth visit based on questionnaire response
Time Frame: Through study completion
Population: Sincere efforts have been made to obtain the results information from the Principal Investigator, but no reportable information has been obtained.
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 0

8. Secondary Outcome: Clinic Savings Derived From Telehealth Visits
Description: Clinic savings derived from telehealth visits v in-person visits
Time Frame: Through study completion
Population: as for outcome 7
Arm/Group | Health Services Research (Telehealth)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: baseline through 16 weeks
Arm/Group | Health Services Research (Telehealth)
All-Cause Mortality (participants affected / at risk) | 2/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT02751580/Prot_SAP_000.pdf